CLINICAL TRIAL: NCT05899907
Title: A Study of Telitacicept in the Treatment of Early Stage Systemic Lupus Erythematosus
Brief Title: Efficacy and Safety of Telitacicept in Early SLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaomei Leng, Principal Investigator, Clinical Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-HS3345D
Record Dates: First submitted 2023-03-26; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus Erythematosus, Systemic; Telitacicept
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Standard of care plus Telitacicept 160 mg sc per week; after week 12, the dose can be reduced to 80 mg per week due to safety considerations.
  Interventions: Drug: Telitacicept; Drug: Standard of Care
- Control group (Other): Standard of care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Telitacicept — 160mg once a week for 48 weeks
  Other Names: RC18
  Arms: Treatment group
Drug: Standard of Care — Steroid(≤1mg/kg/d) with or without proper immunosuppressants：CTX, MMF, AZA, CsA, FK 506, HCQ, MTX, LEF, SASP etc.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Telitacicept in adult patients with early stage of SLE .

DETAILED DESCRIPTION:
This is a phase 4, multicentre, randomised, double-blind, open-labeled study to evaluate the efficacy and safety of telitacicept in adult subjects with active early stage of SLE (disease duration less than 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE according to the 1997 American College of Rheumatology (ACR) classification criteria or 2019 EULAR/ACR classification criteria
* 18-65 years of age
* body weight 45-90kg
* antinuclear antibody titers ≥1:80, and/ or anti-double-stranded DNA antibodies
* SLEDAI-2K score ≥8 scores
* Disease duration less than 2 years (defined as the duration between the first appearance of any symptom/sign attributed to SLE and baseline)
* A stantard therapy for at least 30d for patients who are not treatment-naive
* Negative pregnancy test for child-bearing women at screening and baseline
* Provide written informed consent

Exclusion Criteria:

* Known to be allergic to Prednisone Acetate, Meprednisone, Hydroxychloroquine, and Immunosuppressants including Mycophenolate Mofetil, Cyclophosphamide,et al
* Active serious neuropsychiatric systemic lupus erythematosus or other severe situations of SLE who need pulse steroid treatment
* severe lupus nephritis: 24hUP more than 6g, serum creatinine > 221umol/L
* History of severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis, or CNS vasculitis) requiring intervention within 60 days of baseline (Day 1)
* Abnormal liver function (ALT or AST is 2 times higher than normal)
* Baseline IgG below the lower limit of the normal range
* Pregnancy or breastfeeding women
* Have a history of malignant tumors
* Have any serious acute, chronic or recurrent infectious disease (such as pneumonia or active stage of pyelitis, recurrent pneumonia, chronic bronchiectasis and tuberculosis)
* Chronic infections, such as Hepatitis B virus or hepatitis B and C and HIV
* Cardiac insufficiency with metabolic imbalance or severe high blood pressure (systolic pressure > 160mmHg or diastolic pressure > 100mmHg) or diabetics
* Active hemorrhage or peptic ulcer
* With other concommitant autoimmune disease;
* Receipt of B-cell-targeted therapy (including belimumab) within 1 year before randomization
* Receipt of IVIG within 28 days before randomization
* Receipt of TNF inhibitor, IL-1R inhibitor or plasma exchange therapy within 90 days before randomization
* Participated in other drugs clinical trials within 4 weeks.
* Receipt of live vaccine within 4 weeks before randomization
* Receipt of COVID-19 vaccine within 4 weeks before randomization
* Subjects who in the opinion of the investigator are not suitable to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of LLDAS in week 24 | week 24
  Lupus low disease activity status (LLDAS) was defined as SLEDAI-2K ≤4, no activity in any major organ, no new disease activity feature, PGA ≤1, prednisone ≤7.5 mg/day, and allowance for maintenance of IS and antimalarials

SECONDARY OUTCOMES:
Proportion of LLDAS in week 12 | week 12
  Lupus low disease activity status (LLDAS) was defined as SLEDAI-2K ≤4, no activity in any major organ, no new disease activity feature, PGA ≤1, prednisone ≤7.5 mg/day, and allowance for maintenance of IS and antimalarials
Improvement in SLEDAI-2K | week 24 and 52
  Proportion of patients with SLEDAI-2K scores improvement ≥4 compared with baseline
Improvement in serological indices | week 24, 52
  Improvement in anti-dsDNA antibody titers, C3, C4, T cell and B cell subsets and IgG, IgA, IgM compared with baseline
Change in PGA | week 24, 52
  PGA: physician global assesment(0-3)
Number of participants with Adverse Events | up to week 52
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A SAE is any untoward medical occurrence that at any dose resulting in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant and which the investigator regards as serious based on appropriate medical judgment.
Disease flare | up to week 52
  Proportion of patients suffer from SLE flare

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Leng, Principal Investigator — Peking Union Medical College Hospital
Locations (20):
- China (20):
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing
  - Fuyang People's Hospital, Fuyang
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guanzhou
  - Qilu Hospital of Shandong University, Jinan
  - the First People's Hospital of Yunnan Province, Kunming
  - The Second Affiliated Hospital of Lanzhou University, Lanzhou
  - The Affiliated Hospital of Nantong University, Nantong
  - the Affiliated Hospital of Qingdao University, Qingdao
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Baiqiuen Hospital, Taiyuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - Tongji Hospital, Tongji Medical College,, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuxi Second People's Hospital, Wuxi
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou

IPD SHARING:
Plan to Share IPD: No